CLINICAL TRIAL: NCT03125486
Title: Compassionate Use for Subcutaneous (SC) Belimumab
Status: No longer available | Type: Expanded Access
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207616
Record Dates: First submitted 2017-04-18; First posted 2017-04-24 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: subcutaneous Belimumab; Individual Patient Compassionate Use; SLE; GSK1550188
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: SC belimumab 200 mg — Belimumab subcutaneous 200 mg will be supplied for compassionate use for the identified individual subject.

SUMMARY:
GlaxoSmithKline (GSK) have submitted a Biologic License Application (BLA) for the subcutaneous formulation of belimumab which is currently under review by the Food and Drug Administration (FDA). The goal of this individual patient compassionate use supply is to provide a patient with subcutaneous belimumab for the period of 1 year or until the subcutaneous formulation of belimumab becomes approved for use by the FDA and is commercially available to this patient, whichever is sooner. You can access GSK's Policy on Compassionate via http://www.gsk.com/media/3368/compassionate-use.pdf.

ELIGIBILITY:
This is a protocol to support an emergency IND for compassionate use in one patient requiring use of belimumab subcutaneous for SLE treatment (lacks venous access and cannot receive IV belimumab).

Eligibility criteria is based on the following, as provided within GSK's policy on compassionate use:

* The illness being treated is life threatening or seriously debilitating.
* There are no satisfactory alternative treatments (confirmed by the HCP).
* There is sufficient evidence to believe the benefit to the patient justifies the risk You can access GSK's Policy on Compassionate via http://www.gsk.com/media/3368/compassionate-use.pdf.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Milwaukee, Wisconsin, United States